CLINICAL TRIAL: NCT00828971
Title: A Prospective, Randomized, Open Label, Active Comparator, Multicenter, National Trial to Compare the Efficacy and Safety of Sequential IV/PO Moxifloxacin 400 mg Once Daily Versus IV Amoxicillin/Clavulanate 2,0/0,2 g Every 8 Hours Followed by Oral Amoxicillin/Clavulanate 875/125 mg Every 8 Hours in the Treatment of Adult Subjects With Complicated Skin and Skin Structure Infections
Brief Title: A Study to Assess Efficacy and Safety of IV/PO Moxifloxacin in the Treatment of cSSSIs
Acronym: MERAK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12670; 2007-001491-36 (EudraCT Number)
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Infectious Diseases
Keywords: Complicated skin and skin structure infections; cSSSI
MeSH Terms: conditions — Communicable Diseases | interventions — Moxifloxacin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)
- Arm 2 (Active Comparator)
  Interventions: Drug: Amoxicilline/clavulanic

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Sequential IV/PO moxifloxacin 400/400 mg every 24 hours, for 7 to 21 days.
  Arms: Arm 1
Drug: Amoxicilline/clavulanic — IV Amoxicilline/clavulanic acid 2000/200 mg TID followed by PO amoxicilline/clavulanate 875/125 mg TID for a total of 7 to 21 days
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess if a therapy with intravenous and oral moxifloxacin is as effective as a therapy with intravenous and oral amoxicilline/clavulanate in the treatment of complicated skin and skin structure infection.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Men or women of age >/= 18 years with a diagnosis of bacterial skin and skin structure infection that requires

  * Hospitalization
  * Initial parenteral therapy for at least 48 hours
* Complicated by at least one of the following criteria:

  * Involvement of deep soft tissues (e.g. fascial, muscle layers)
  * Requirement for a significant surgical intervention including surgical drainage, drainage procedure guided by imaging and/or debridement
  * Association with a significant underlying disease that may complicate response to treatment.
  * Presence of SIRS (Systemic Inflammatory Response Syndrome) defined as two or more of the following signs or symptoms: - temperature > 38.3°C or < 36°C - white blood cell count > 12.000/mmc or < 4.000 or > 10% bands - pulse rate > 90 beats/min - respiratory rate > 20178 - systolic blood pressure </= 90 mmgHg - decreased capillary refill/mottling > 2 seconds - lactate > 2 mmol/L - altered mental status - hyperglycemia > 120 mg/dl or 7.7 mmol/L in the absence of diabetes - protein C (CPR) > 20 mg/L (VR 0-5)3. Duration of infection < 21 days
* Diagnosis of one of the following skin and skin structure infections:

  * major abscess(es) associates with extensive cellulitis
  * erysipelas and cellulitis
  * infected pressure ulcers(s)
  * wound infections including: post surgical (surgical incision), post traumatic, human bite/clenched fist and animal bite wound and wound associated with injection drug abuse
  * Infected ischemic ulcers with at least one of the following conditions: - Diabetes mellitus - Peripheral vascular disease - Conditions pre-disposing to pressure scores such as paraplegia or peripheral neuropathy
* Presence of at least 3 of the following local signs and symptoms

  * purulent drainage or discharge
  * erythema extended >1 cm from the wound edge
  * fluctuance
  * pain or tenderness to palpation
  * swelling or induration
  * fever defined as body temperature > 37.5°C (axillary), > 38°C (orally), > 38.5°C (tympanically), or > 39°C (rectally). OR Elevated total peripheral white blood cell (WBC) count> 12,000/mm3 OR > 15% immature neutrophils (blends) regardless of total peripheral WBC count
  * C-reactive protein (CRP) >20 mg/L

Exclusion Criteria:

* Women, who are pregnant or lactating, or in whom pregnancy can not be excluded (Note: a urine pregnancy test has to be performed for all women of childbearing potential before randomization to the study drug).
* The following skin and skin structure infections:

  * Necrotizing fasciitis including Fournier's gangrene, ecthyma gangrenosum, streptococcal necrotizing fasciitis and clostridial necrotizing fasciitis.
  * Burn wound infections.
  * Secondary infections of a chronic skin disease (eg, atopic dermatitis).
  * Infection of prosthetic materials. Subjects with removal of a prosthetic device involved in an infection should not be included.
  * Infections where a surgical procedure alone is definitive therapy.
  * Subjects with uncomplicated skin and skin structure infections including

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Clinical response up to 14-21 days after the completion of study drug therapy (Test-of-Cure visit [TOC]). | Test-of-Cure visit [TOC].

SECONDARY OUTCOMES:
Clinical response assessed by the investigator on treatment Day 3-5 | Day 3-5
Clinical response assessed by the investigator at the end-of-therapy (EOT). | At the end-of-therapy (EOT)
Time to switch from oral to IV therapy | Day of switch from oral to IV therapy
Bacteriological response (for microbiologically valid population) at the EOT and TOC | At the end-of-therapy (EOT), Test-of-Cure visit [TOC].

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- Italy (21):
  - Bagno Di Ripoli, Firenze
  - Bari
  - Bergamo
  - Bologna
  - Brescia
  - Ferrara
  - Florence
  - Foggia
  - Genova
  - Mantova
  - Messina
  - Napoli
  - Padua
  - Perugia
  - Reggio Emilia
  - Rimini
  - Roma
  - Torino
  - Udine
  - Varese
  - Verona

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/